CLINICAL TRIAL: NCT07215364
Title: Impact of EXercise on Quality of Life of Early Breast Cancer Patients on Treatment With Adjuvant Aromatase Inhibitors With or Without CDK4/6 Inhibitors. "The EXAI Study"
Brief Title: Impact of Exercise on Quality of Life of EBC Patients on Treatment With Adjuvant AI With or Without CDK4/6 Inhibitors
Acronym: EX-AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GEICAM/2023-09; 2025-522848-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-01; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Early-stage Breast Cancer
Keywords: early-stage breast cancer (EBC); HR-positive; HER2-negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Approximately 37 patients in the experimental group will perform a 6-month training program consisting of exercise sessions 3 alternating days per week (combined resistance + aerobic exercise).
  Interventions: Behavioral: Training program
- Control group (No Intervention): Approximately 37 patients in the control group will receive usual health care. This patients' group will be provided with the international exercise guidelines for cancer patients.

INTERVENTIONS:
Behavioral: Training program — Training program consist on physical activity sessions (combined resistance plus aerobic exercises) that will be performed 3 times per week every-other-day.
  Arms: Experimental group

SUMMARY:
This is a national clinical trial (Spain), conducted in approximately 5 sites, where patients who agree to participate will be included in one of two exercise program groups: the experimental group (a combined resistance and aerobic exercise program) and the control group.

The study will begin with a pilot phase involving approximately 74 patients.

Approximately 37 patients in the experimental group will follow a 6-month training program consisting of exercise sessions three alternate days per week (combining resistance and aerobic exercise).

Approximately 37 patients in the control group will receive standard medical care. These patients will be provided with international exercise guidelines for cancer patients.

Patients will continue with their assigned physical activity intervention until the maximum number of months for the intervention, unacceptable toxicity, discontinuation of hormone therapy, or withdrawal of consent-whichever occurs first.

DETAILED DESCRIPTION:
Study population:

The target population for randomization in this study includes women diagnosed with Hormone receptor (HR)+/Human epidermal growth factor receptor 2 (HER2)-negative- early-stage breast cancer (EBC) and who have already received between 10 and 18 weeks of an AI (with or without a LHRHa) before the randomization in the study. Those patients that are candidates to receive an adjuvant CDK4/6i should have initiated the treatment at least 6 weeks before the randomization in the study.

Study treatment:

Although patients should receive adjuvant ET (including an AI [steroidal inhibitors such as exemestane or non-steroidal inhibitors such as anastrozole or letrozole], with or without a CDK4/6i and with or without a LHRHa) to be eligible for this study, the clinical decisions concerning the optimum management strategy for a particular patient will be taken independently of and prior to any decision by the investigator to invite a patient to participate in the study and according to the approved product information, local treatment guidelines and/or routine clinical practice.

The EX-AI study has been developed to be pragmatic as it adheres to local guidelines for the use of ET in the adjuvant setting. There are no extra tests or assessments required as we allow patients management to follow the standard of care. The burden on patients is limited to completing the training program and questionnaires/scales. The diagnostic and monitoring procedures used do not introduce any risk or burden beyond those associated with routine clinical practice in Spain.

The study is mainly focused on the completion of physical activity interventions by patients and its effect on their QoL rather than the adjuvant treatment that they will be receiving.

Study duration:

The study start date is the date of the first site activation. It is estimated that the accrual will be completed in approximately 18 months. The end of study (EoS) date is the date of the last visit of the last patient (LPLV =last patient last visit), considering 6 months of the exercise program, and its potential extension for 6 additional months depending on the progress of the study and once the necessary funding for this extension has been obtained; in case it is extended, patients in both groups will be able to choose whether they would want to continue in the study for these additional 6 months follow-up. If the patients in the control group agree to continue, then they would have a passive follow-up (i.e., maintaining the same physical activity that they performed up to date). The patients in the experimental group that agree to continue would be able to choose to continue in the study through an active or passive follow-up; if they decide to continue in an active follow-up, then they would continue with the training program as previously performed; if they choose to continue in the passive follow-up on the contrary, then they would not continue with the training program as previously performed but would be encouraged to remain physically active considering international recommendations (like in the control group).The evaluation of the exploratory objectives will be independent of the EoS date.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent document (ICD) prior to any specific study procedures, showing patience, willingness and ability to comply with the physical activity program in the experimental group, and scheduled visits and study procedures in both groups.
2. Patients ≥18 years of age at signing of ICD.
3. Documented histologically confirmed HR+/HER2- invasive EBC, adequately treated according to standard clinical practice and with absence of any evidence of disease (loco-regional or metastatic at distance).

   HR and HER2 assessments are performed under institutional guidelines.
   * HR testing should utilize an assay consistent with the most recent American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) Guidelines.
   * HER2 negativity is determined as immunohistochemistry (IHC) score 0/1+ or negative by in situ hybridization (ISH) according to the recommendations of the most recent ASCO/CAP Guidelines.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
5. Pre-, peri-, and post-menopausal women (as determined by the investigator and according to the institutional guidelines) that have already received between 10 and 18 weeks of an AI (with or without a LHRHa) before the randomization in the study and administered according to local guidelines.

   Note: Patients that are candidate to receive an adjuvant CDK4/6i will only be eligible if the CDK4/6i was initiated at least 6 weeks before the randomization in the study and administered according to local guidelines.
6. Patients must have undergone adequate (definitive) loco-regional therapy (surgery with or without radiation therapy), with or without neo-/adjuvant systemic CT.
7. Patients must have an adequate organ and bone marrow function according to the standard clinical practice and institutional guidelines.
8. Patients must be able and willing to fill out repeated questionnaires on QoL, pain and fatigue, as well as to adhere to the physical activity program.
9. Fluent Spanish language skills for the complete comprehension of the questionnaires.
10. With the consent of the investigator for participation in physical training and considering the medical history of the patient.

Exclusion Criteria:

1. Patients have received less than 10 weeks or more than 18 weeks of an AI (with or without a LHRHa) before the randomization in the study.
2. Patients that are candidate to receive an adjuvant CDK4/6i initiated the treatment less than 6 weeks before the randomization in the study.
3. Patients have musculoskeletal injuries.
4. Patients have known significant heart disease (myocardial infarction, unstable angina, congestive heart failure, cardiomyopathy, etc.).
5. Patients with weight over 150kg.
6. Patients have any type of illness or mental condition that prevents or compromises the well-being of the patient or compliance with the procedures.
7. Patients have any cardiovascular contraindication to physical training by the investigator.
8. Patients have been performing supervised training, either aerobic and/or resistance training (at a gym [group or individual classes] or in a specific sport), at least 2 days per week in the past 6 months.
9. No access and/or unable to manage the website and other digital tools (i.e. applications) for training sessions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Effect of a training program in quality of life questionnaire (QoL)-related to endocrine therapy | Through study treatment, and average of 12 months
  To determine the changes from baseline in the QoL-related to endocrine therapy (ET) symptoms measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer 45 (EORTC QLQ-BR45) questionnaire (questions 54-56, 63-69).
  To calculate the scores for each desirable dimension Scoring Manuals will be followed. Summary statistics (mean, mean confidence interval (CI), standard deviation, median and range) of absolute scores and their changes from baseline will be summarized at each assessment time. The comparison between treatment groups will be performed using a linear mixed model.
  Patients will complete this questionnaire at at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.

SECONDARY OUTCOMES:
Change from baseline in global QoL | Through study treatment, and average of 12 months
  It will be evaluated by the EORTC QLQ-C30 questionnaire (questions 29 and 30). The questionnaire employs twenty-eight 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QoL. For functional and global QoL scales, higher scores represent a better level of functioning and are converted to a 0 to 100 scale. For symptom-oriented scales, a higher score represents more severe symptoms.
  To calculate the scores for each desirable dimension Scoring Manuals will be followed. Summary statistics (mean, mean CI, standard deviation, median and range) of absolute scores and their changes from baseline will be summarized at each assessment time. The comparison between treatment groups will be performed using a linear mixed model.
  Patients will complete this questionnaire at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.
Aromatase inhibitor associated musculoskeletal syndrome (AIMSS) | Through study treatment, and average of 12 months
  AIMSS will be assessed using the Brief Pain Inventory (BPI) scale. The BPI is a 14-item questionnaire developed for cancer patients to assess the worst pain, pain severity, and pain interference over the past week, reported on a scale of 0 to10. Worst pain is categorized as mild (score from 3 to 4), moderate (score from 5 to 7), or severe pain (score from 8 to 10). Pain severity is measured as the average of responses to questions on worst pain, average pain, least pain, and pain right now. Pain interference is the average of 7 interference items, such as walking, mood, and sleep. The BPI is the most common, valid, and reliable measure to assess joint pain in cancer survivors.
  Patients will complete this scale at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.
Fatigue | Through study treatment, and average of 12 months
  Fatigue will be measured by the Brief Fatigue Inventory (BFI) scale, which is a one-dimensional questionnaire based on the Brief Pain Inventory (BPI) that assesses the severity and impact of oncologic pain. The BFI is a scale with 11 points (0 to 10), including a dichotomous question about whether the patient felt tired or fatigued in the last 7 days. For each question, 0 is considered "no fatigue" and 10 is "worst fatigue possible," except for the dichotomous question that is not scored.
  Among the other questions, 3 measures the severity of fatigue in the current, daily situations, and in the last 24 hours. Six questions measure the influence of fatigue in general activities.
  The total score is the average of all questions. According to the total score, fatigue is classified as mild (from 1 to 3 points), moderate (from 4 to 6 points), and severe (from 7 to 10 points).
  Patients will complete this scale at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.
Compliance to treatment | Through study treatment, and average of 12 months
  Compliance to treatment will be recorded using the pill counting method and patient diary.
  Drug compliance is defined as the percentage of doses a study participant has taken (actual consumed dose) compared to the total number of doses prescribed by their physician. The prescribed total dose refers to the comprehensive quantity of medication that is intended to be administered to a patient over a designated treatment period.
Body composition | Through study treatment, and average of 12 months
  Body composition will be measured by bioimpedance scale, which provides information about body composition. This test is performed with special scales (Tanita® or Omron®) which have metal plates to conduct a very low-intensity electric current that travels through the lower limbs, allowing for the assessment of their resistance. These scales show the amount of lean, muscle, and fat mass, water percentage, bone density, and basal metabolic rate based on sex, age, height, and the intensity of physical activity.
  Resistance depends on the amount of water present in the body, with a constant proportion in muscle mass. By relating this data to other factors such as age, sex, and height, muscle mass can be calculated.
  Fat mass = weight - muscle mass. This method considers all the fat in the body, including localized fat, with a margin of error of 3-5%.
Adherence to the physical activity program | Through study treatment, and average of 12 months
  Adherence to the physical activity program will be recorded through the physical exercise professionals' assistance and assessment and through the virtual training platform "10 Mets".
Information on sexual relations: libido | Through study treatment, and average of 12 months
  Libido will be evaluated through the specific questions 44, 45 and 46 included in the EORTC QLQ-BR45 questionnaire.
  To calculate the scores for each desirable dimension Scoring Manuals will be followed. Summary statistics (mean, mean CI, standard deviation, median and range) of absolute scores and their changes from baseline will be summarized at each assessment time. The comparison between treatment groups will be performed using a linear mixed model.
  Patients will complete this questionnaire at at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.
Information on sexual relations: body image | Through study treatment, and average of 12 months
  Body image will be evaluated through the specific questions 39, 40, 41 and 42 included in the EORTC QLQ-BR45 questionnaire.
  To calculate the scores for each desirable dimension Scoring Manuals will be followed. Summary statistics (mean, mean CI, standard deviation, median and range) of absolute scores and their changes from baseline will be summarized at each assessment time. The comparison between treatment groups will be performed using a linear mixed model.
  Patients will complete this questionnaire at at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.
Information on sexual relations: vaginal dryness | Through study treatment, and average of 12 months
  Vaginal dryness will be evaluated through the specific questions 70, 71, 72 and 73 included in the EORTC QLQ-BR45 questionnaire.
  To calculate the scores for each desirable dimension Scoring Manuals will be followed. Summary statistics (mean, mean CI, standard deviation, median and range) of absolute scores and their changes from baseline will be summarized at each assessment time. The comparison between treatment groups will be performed using a linear mixed model.
  Patients will complete this questionnaire at at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.
Cognitive impairment | Through study treatment, and average of 12 months
  Cognitive impairment will be evaluated through the specific questions 20 and 25 included in the EORTC QLQ-C30 questionnaire.
  To calculate the scores for each desirable dimension Scoring Manuals will be followed. Summary statistics (mean, mean CI, standard deviation, median and range) of absolute scores and their changes from baseline will be summarized at each assessment time. The comparison between treatment groups will be performed using a linear mixed model.
  Patients will complete this questionnaire at at baseline and during physical activity intervention: 1.5, 3, 6 and 12 months.
The Number of Participants Who Experienced Adverse Events (AE) Related to Study Treatment | Through study treatment, and average of 12 months
  Safety assessments will be performed at baseline and during the study: Vital signs assessments (blood pressure, pulse and body temperature), triplicate 12-lead electrocardiogram (as clinically indicated), laboratory assessments (Hemoglobin, white blood cells count, absolute neutrophils count, lymphocytes, platelets count, glucose, alkaline phosphatase, gamma glutamyl transferase, alanine aminotransferase, aspartate aminotransferase, total bilirubin, serum creatinine, sodium, potassium, cholesterol, triglycerides, uric acid, BUN), pregnancy test (as clinically indicated).
  AE grade will be defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 5.0.
  Safety will be assessed by the incidence of AEs by maximum grade of severity of NCI CTCAE version 5.0.
Tolerability to the treatment | Through study treatment, and average of 12 months
  Tolerability will be assessed by incidence of treatment dose modifications, discontinuations due to AEs, number of administered cycles, dose intensity, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Universitario Clínico San Cecilio, Granada, Spain; Study Director, Study Director — Hospital Quirón Sagrado Corazón-Sevilla, Sevilla, Spain
Locations (5):
- Spain (5):
  - Institut Català d'Oncología (ICO) L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quirón Sagrado Corazón de Sevilla, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Multidisciplinary academic group leading in breast cancer research, education, and patient support — http://www.geicam.org